CLINICAL TRIAL: NCT04017156
Title: Bone Healing at Non-submerged Implants Installed With Different Insertion Torques. A Split Mouth Histomorphometric Randomized Controlled Trial.
Brief Title: Bone Healing at Non-submerged Implants Installed With Different Insertion Torques.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARDEC Academy (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: protocol #04-2014
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Edentulous; Alveolar Process, Atrophy
MeSH Terms: conditions — Mouth, Edentulous; Atrophy

STUDY DESIGN:
Intervention Model Description: Clinical Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The two recipient sites will be selected prior the surgery, while the type of site preparation will be randomly decided. The randomization will be performed electronically (randomization.com) by a researcher neither involved in the selection of the patients nor in installation of the devices (DB). Sealed opaque envelopes will be prepared and opened at the time of surgery by an author not involved in the surgery (DB). Surgeon and patients will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test site (torque of <10 Ncm) (Experimental): The test sites (<10 Ncm) will be over-prepared with drills of larger diameter
  Interventions: Procedure: implant installation
- Control site (torque of ~30 Ncm) (Other): the standard sites (~30 Ncm)will be prepared with the corresponding drills suggested by the manufacturer
  Interventions: Procedure: implant installation

INTERVENTIONS:
Procedure: implant installation — All site preparations will be performed deeper compared to the length of the implant so that the implant apex cannot reach the bottom of the osteotomy.
  Other Names: implant surgery

SUMMARY:
The objective of the study is to evaluate histomorphometrically the healing at implants installed with standard or very low insertion torque values.

DETAILED DESCRIPTION:
Very high insertion torque values have been recommended when immediate loading is applied to implants.1 However, it has been shown that similar clinical outcomes may be achieved even with insertion torque values ≤15 Ncm when implants are splinted together. Due to the contradictory outcomes on the influence of the torque on osseointegration and a lack of histological data in humans, there is a need of more evidences that may support the clinicians in the decision making when an unintentional low insertion torque occur at implants during the daily practice. So the aim of the study i evaluate histomorphometrically the healing at implants installed in Twelve volunteer patients that will be recruited. Two screw-shaped titanium devices will be installed in the distal segments of the mandible using insertion torque values of either <10 Ncm or ~30 Ncm. The implants were left to heal in a non-submerged fashion. After 8 weeks, biopsies will be retrieved and ground sections will be prepared for histological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least two edentulous zone in the posterior segment of the mandible
* ≥ 25 years of age
* smoking ≤ 10 cigarettes per day
* Good general health
* No contraindication for oral surgical procedures.
* Not being pregnant.

Exclusion Criteria:

* Presence of systemic disorders
* Chemotherapy or radiotherapy;
* Smokers >10 cigarettes per day
* Previous bone augmentation procedures in the region

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
New bone in contact with the implant surface | After 8 weeks of healing
  The percentages of new bone will be evaluated both in contact with the implant surface

SECONDARY OUTCOMES:
Bone density around the implant surface | After 8 weeks of healing
  The total mineralized bone will be assessed as sum of new and old bone

OTHER OUTCOMES:
pre-existing (old) bone, soft tissue (marrow spaces, Haversian canals, BMUs canals), bone debris/ clot remnants, and marrow spaces (soft tissue) | After 8 weeks of healing
  The percentages of pre-existing (old) bone, soft tissue (marrow spaces, Haversian canals, BMUs canals), bone debris/ clot remnants, and marrow spaces (soft tissue) will be evaluated all in contact with the implant surface

CONTACTS AND LOCATIONS:
Locations (1):
- Colombia, Cartagena, Cartagena, Colombia

IPD SHARING:
Plan to Share IPD: No
Will be shared after publication

REFERENCES:
- [Result] Trisi P, Todisco M, Consolo U, Travaglini D. High versus low implant insertion torque: a histologic, histomorphometric, and biomechanical study in the sheep mandible. Int J Oral Maxillofac Implants. 2011 Jul-Aug;26(4):837-49. PMID 21841994
- [Result] Cesaretti G, Botticelli D, Renzi A, Rossi M, Rossi R, Lang NP. Radiographic evaluation of immediately loaded implants supporting 2-3 units fixed bridges in the posterior maxilla: a 3-year follow-up prospective randomized controlled multicenter clinical study. Clin Oral Implants Res. 2016 Apr;27(4):399-405. doi: 10.1111/clr.12565. Epub 2015 Feb 9. PMID 25664701
- [Result] Gallucci GO, Benic GI, Eckert SE, Papaspyridakos P, Schimmel M, Schrott A, Weber HP. Consensus statements and clinical recommendations for implant loading protocols. Int J Oral Maxillofac Implants. 2014;29 Suppl:287-90. doi: 10.11607/jomi.2013.g4. No abstract available. PMID 24660204
- [Result] Pantani F, Botticelli D, Garcia IR Jr, Salata LA, Borges GJ, Lang NP. Influence of lateral pressure to the implant bed on osseointegration: an experimental study in dogs. Clin Oral Implants Res. 2010 Nov;21(11):1264-70. doi: 10.1111/j.1600-0501.2010.01941.x. PMID 20626423
- [Result] Rea M, Lang NP, Ricci S, Mintrone F, Gonzalez Gonzalez G, Botticelli D. Healing of implants installed in over- or under-prepared sites--an experimental study in dogs. Clin Oral Implants Res. 2015 Apr;26(4):442-446. doi: 10.1111/clr.12390. Epub 2014 Mar 31. PMID 24684411
- [Result] Rea M, Botticelli D, Ricci S, Soldini C, Gonzalez GG, Lang NP. Influence of immediate loading on healing of implants installed with different insertion torques--an experimental study in dogs. Clin Oral Implants Res. 2015;26(1):90-5. doi: 10.1111/clr.12305. Epub 2013 Dec 9. PMID 24313303
- [Result] Barone A, Alfonsi F, Derchi G, Tonelli P, Toti P, Marchionni S, Covani U. The Effect of Insertion Torque on the Clinical Outcome of Single Implants: A Randomized Clinical Trial. Clin Implant Dent Relat Res. 2016 Jun;18(3):588-600. doi: 10.1111/cid.12337. Epub 2015 Jun 5. PMID 26043651
- [Result] Verardi S, Swoboda J, Rebaudi F, Rebaudi A. Osteointegration of Tissue-Level Implants With Very Low Insertion Torque in Soft Bone: A Clinical Study on SLA Surface Treatment. Implant Dent. 2018 Feb;27(1):5-9. doi: 10.1097/ID.0000000000000714. PMID 29271785
- [Result] Verrastro Neto A, Andrade R, Correa MG, Casarin RCV, Casati MZ, Pimentel SP, Ribeiro FV, Cirano FR. The impact of different torques for the insertion of immediately loaded implants on the peri-implant levels of angiogenesis- and bone-related markers. Int J Oral Maxillofac Surg. 2018 May;47(5):651-657. doi: 10.1016/j.ijom.2017.11.001. Epub 2017 Nov 23. PMID 29173997
- [Result] Duyck J, Corpas L, Vermeiren S, Ogawa T, Quirynen M, Vandamme K, Jacobs R, Naert I. Histological, histomorphometrical, and radiological evaluation of an experimental implant design with a high insertion torque. Clin Oral Implants Res. 2010 Aug;21(8):877-84. doi: 10.1111/j.1600-0501.2010.01895.x. Epub 2010 Apr 30. PMID 20528892
- [Result] Duyck J, Roesems R, Cardoso MV, Ogawa T, De Villa Camargos G, Vandamme K. Effect of insertion torque on titanium implant osseointegration: an animal experimental study. Clin Oral Implants Res. 2015 Feb;26(2):191-6. doi: 10.1111/clr.12316. Epub 2013 Dec 11. PMID 24325598
- [Result] Muktadar AK, Gangaiah M, Chrcanovic BR, Chowdhary R. Evaluation of the effect of self-cutting and nonself-cutting thread designed implant with different thread depth on variable insertion torques: An histomorphometric analysis in rabbits. Clin Implant Dent Relat Res. 2018 Aug;20(4):507-514. doi: 10.1111/cid.12611. Epub 2018 Apr 16. PMID 29659124
- [Result] Berardini M, Trisi P, Sinjari B, Rutjes AW, Caputi S. The Effects of High Insertion Torque Versus Low Insertion Torque on Marginal Bone Resorption and Implant Failure Rates: A Systematic Review With Meta-Analyses. Implant Dent. 2016 Aug;25(4):532-40. doi: 10.1097/ID.0000000000000422. PMID 27129002
- [Result] Balshi SF, Wolfinger GJ, Balshi TJ. A retrospective analysis of 44 implants with no rotational primary stability used for fixed prosthesis anchorage. Int J Oral Maxillofac Implants. 2007 May-Jun;22(3):467-71. PMID 17622014
- [Result] Rodrigo D, Aracil L, Martin C, Sanz M. Diagnosis of implant stability and its impact on implant survival: a prospective case series study. Clin Oral Implants Res. 2010 Mar;21(3):255-61. doi: 10.1111/j.1600-0501.2009.01820.x. Epub 2009 Dec 4. PMID 19958375
- [Result] Caneva M, Lang NP, Calvo Guirado JL, Spriano S, Iezzi G, Botticelli D. Bone healing at bicortically installed implants with different surface configurations. An experimental study in rabbits. Clin Oral Implants Res. 2015 Mar;26(3):293-9. doi: 10.1111/clr.12475. Epub 2014 Sep 15. PMID 25220835
- [Result] Ferri M, Lang NP, Angarita Alfonso EE, Bedoya Quintero ID, Burgos EM, Botticelli D. Use of sonic instruments for implant biopsy retrieval. Clin Oral Implants Res. 2015 Nov;26(11):1237-43. doi: 10.1111/clr.12466. Epub 2014 Aug 11. PMID 25109369
- [Derived] Amari Y, Piattelli A, Apaza Alccayhuaman KA, Mesa NF, Ferri M, Iezzi G, Botticelli D. Bone healing at non-submerged implants installed with different insertion torques: a split-mouth histomorphometric randomized controlled trial. Int J Implant Dent. 2019 Dec 5;5(1):39. doi: 10.1186/s40729-019-0194-2. PMID 31802302

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT04017156/Prot_SAP_000.pdf